CLINICAL TRIAL: NCT02826889
Title: Assessing the Diagnostic Accuracy of Corrected Flow Time (FTc) and Pleth Variability Index (PVI) as Predictors of Fluid Responsiveness in Patients in the Prone Position Using the Jackson Table
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2016-0189
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Elective Posterior Lumbar Spinal Fusion for Spinal Stenosis; Spondylolisthesis; Spinal Fractures; Scoliosis or Tumors
Keywords: Fluid responsiveness; corrected flow time; pleth variability index; prone position
MeSH Terms: conditions — Spondylolisthesis; Spinal Fractures; Scoliosis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluid loading group (Experimental)
  Interventions: Device: Philips Intelivue MP70 monitor; Device: Pleth Variability Index (PVI)

INTERVENTIONS:
Device: Philips Intelivue MP70 monitor — Philips Intelivue MP70 monitor (Intellivue MP70, Philips medical Systems, Suresnes, France) -a radial arterial cannula is inserted and arterial pressure waveforms are monitored through Philips Intelivue MP70 monitor. In the monitor, PPVauto is displayed in real-time. It is based on automatic detection algorithms, kernel smoothing, and rank-order filters.
Device: Pleth Variability Index (PVI) — PVI is the measure of the dynamic changes in the Perfusion Index (PI) that occur during one or more complete respiratory cycles. A rainbow Pulse CO-Oximetry sensor is attached to the patient's finger and the PVI is displayed in real-time on the Root monitor.

SUMMARY:
Appropriate fluid management is an important part of anesthesia in patients undergoing surgery, and several dynamic indices have been suggested to have high predictability for fluid responsiveness in patients receiving mechanical ventilation. Among various surgical positions, the prone position is known to cause unique physiologic and hemodynamic changes and affect the predictability and cut-off values of dynamic indices for fluid responsiveness. A previous study reported that pulse pressure variation (PPV) and corrected flow time were able to predict fluid responsiveness with relatively high accuracy in patients undergoing spine surgery in the prone position using a Wilson frame. However, the Jackson frame is known to have less effects on the cardiovascular system compared to the Wilson frame, and therefore may be physiologically more appropriate in patients undergoing surgery in the prone position. The pleth variability index (PVI) is a dynamic index that can be monitored non-invasively in patients under mechanical ventilation. The present study aims evaluate the validity of PPV and pleth variability index (PVI) as predictors of fluid responsiveness in the supine and prone positions in patients undergoing posterior lumbar spinal fusion using the Jackson table.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the age of 19 and 75, scheduled for spine surgery under general anesthesia using the Jackson table

Exclusion Criteria:

1. Patient refusal
2. Patients that are not normal sinus rhythm on preoperative ECG
3. Patients with moderate~severe cardiac valve disease
4. Patients with an ejection fraction under 50%
5. Significant lung disease
6. Obesity (BMI>35kg/m2)
7. Patients with contraindications to esophageal doppler probe insertion
8. Illiterate patients or foreigners

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Pulse Pressure Variation (PPV) | From 15 minutes after induction of anesthesia in the supine position to 5 minutes after fluid loading in the prone position
  Fluid responsiveness predictability of FTc and PVI in patients undergoing posterior lumbar fusion in the prone position by using the Jackson frame by calculating area under the curve of the ROC curve.
Pleth Variability Index (PVI) | From 15 minutes after induction of anesthesia in the supine position to 5 minutes after fluid loading in the prone position

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea